CLINICAL TRIAL: NCT04595110
Title: Extensive Investigation of the Hemostatic Profile in a Prospective Cohort of Patients Affected by COVID-19
Brief Title: Hemostatic Profile in Patients Affected by COVID-19
Acronym: EMO-COVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ANNA FALANGA (Other)
Responsible Party: Sponsor-Investigator, ANNA FALANGA, Principal Investigator, A.O. Ospedale Papa Giovanni XXIII
Organization: A.O. Ospedale Papa Giovanni XXIII (Other)
Other Study IDs: EMO-COVID-ASSTPG23
Record Dates: First submitted 2020-09-14; First posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Covid19; Thrombosis
Keywords: covid19; Hospitalized patients; coagulation
MeSH Terms: conditions — COVID-19; Thrombosis | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for hemostasis study are collected from all study subjects at admission. After discarding the first 2-3 mL of blood, peripheral venous blood samples were collected into 6 mL vacuum tubes (BD, Vacutainer ™, Plymouth, UK) containing 3.2% citrate (0.109 mol/L, 1:9 vol./vol.) for coagulation studies, and K3-ethylenediamine tetraacetic acid (K3-EDTA) 7.2mg for the complete blood cell count study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational study — Coagulation factors, Hypercoagulation biomarkers, Endothelial, Fibrinolysis and neutrophil activation biomarkers

SUMMARY:
Coronavirus disease-2019 (COVID-19), a viral respiratory illness caused by the severe acute respiratory syndrome-coronavirus-2 (SARS-CoV-2), has been associated with the occurrence of cardiovascular adverse events including acute myocardial injury, acute heart failure, cardiac arrhythmias, and thromboembolic disease. These complications represent an important issue in COVID-19 patients accounting for the increased morbidity and mortality of this syndrome. According to a scoping review, venous thromboembolism and stroke occurred in approximately 20% and 3% of patients, respectively, with higher frequency observed in severely ill patients admitted to intensive care units. Despite the use of pharmacological thromboprophylaxis, the thrombotic risk still remained elevated in severe COVID-19 patients, and the optimal doses and timing of anticoagulation are not yet defined. The pathogenesis of COVID-19 associated thrombosis recognizes a prominent role of endothelial damage induced by both direct viral injury and an excessive and aberrant hyper-inflammatory host immune response associated to an increase in infection-related cytokines and chemokines. The occurrence of a hypercoagulable state in COVID-19 patients associated to a profound endothelial cell activation/dysfunction can result in the pathological phenomenon of immunothrombosis.

In this study, in a prospective cohort of consecutive COVID-19 hospitalized patients, an extensive characterization of the hemostatic alterations were performed, in order to: 1) clarify mechanisms underlying the coagulopathy in these patients; 2) how and to what extent the concomitant infection with SARS-CoV-2 affect this coagulopathy; and 3) identify biomarkers potentially predictive of disease outcome (i.e. any thrombotic recurrence and death).

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* Adult patients admitted with severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) positivity (by real time-PCR) from nasal swab or deep respiratory specimen or with clinical signs suggestive of SARS-Cov-2
* Patients who have signed informed consent. If there is no possibility of obtaining informed consent for the clinical picture (eg adult patients sedated and curarized for acute respiratory failure and consequent mechanical ventilation), the patient's consent will be assumed until the contrary will be manifested.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study involves the enrollment of ≥ 400 consecutive hospitalized patients diagnosed with COVID-19, aged> 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-03-25 (Actual); Primary Completion 2021-04-25 (Estimated); Study Completion 2021-05-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of mortality among enrolled COVID-19 patients | up to 6 months from the date of the enrollment
  Identification of variables for prediction of mortality derived from review of clinical records. Samples collected from identified participants with COVID19 diagnosis will be assessed to determine thrombotic and inflammatory biomarkers able to prediction of mortality.
Incidence of thrombosis among enrolled COVID patients | up to 12 months from the date of the enrollment
  Identification of COVID-19 patients with evidence of thrombotic event derived from review of clinical records. Samples collected from identified participants with COVID19 diagnosis will be assessed to determine thrombotic and inflammatory biomarkers.

SECONDARY OUTCOMES:
Evaluation the role of enoxaparin in the management of Covid-19-associated coagulopathy | Samples collected from identified participants with COVID19 diagnosis will be assessed to determine the effect of thromboprophylaxis on thrombotic and inflammatory biomarkers
  up to 12 months from the date of the enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Papa Giovanni XXIII Hospital - S.I.M.T., Bergamo, Italy

IPD SHARING:
Plan to Share IPD: No